CLINICAL TRIAL: NCT06041815
Title: A Prospective and Observational Clinical Study of the Correlation Between Gut Microbiota and Clinical Response to CAR-T Treatment for Hematological Malignancies
Brief Title: Correlation Between Gut Microbiota and Clinical Response to CAR-T Treatment for Hematological Malignancies
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: The First Affiliated Hospital of Soochow University (Other)
Responsible Party: Sponsor
Other Study IDs: gut microbiota + CAR-T
Record Dates: First submitted 2023-09-11; First posted 2023-09-18 (Actual); Last update posted 2023-09-18 (Actual); Status verified 2023-09

CONDITIONS: Hematological Malignancies; Chimeric Antigen Receptor T-cell Therapy
Keywords: gut microbiota, CAR-T
MeSH Terms: conditions — Hematologic Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — feces
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The purpose of this prospective and observational study is to evaluate the correlation between gut microbiota and clinical response to CAR-T treatment for hematological malignancies

DETAILED DESCRIPTION:
Chimeric antigen receptor T-cell (CAR-T) therapy has shown impressive efficacy in hematological malignancies. However, response rates and associated immune-related adverse effects widely vary among patients. And no biomarkers have been identified to predict the efficacy and associated toxicities after CAR-T therapy in patients. Several preclinical experiments and clinical studies have shown that gut microbiota was associated with the efficacy of T cell-driven cancer immunotherapies and their toxicities. In hematologic malignancies, gut microbiota was associated with the development of graft-versus-host disease (GVHD) after allogeneic hematopoietic stem cell transplantation (allo-HSCT). However, the potential correlation between gut microbiota and the effificacy and toxicity of CAR-T therapy is unclear. Therefore, in this study, we aim to evaluate the correlation between gut microbiota and clinical response to CAR-T treatment for hematological malignancies.

ELIGIBILITY:
Inclusion Criteria:

1. Age 16-65 years.
2. Hematologic malignancies intended for CAR-T therapy.
3. Expected survival time ≥ 3 months (according to investigator's judgement).
4. Left ventricular ejection fractions ≥ 55% by echocardiography.
5. ALT / AST <3 times of normal amounts.
6. Creatinine<2.0mg/dl.
7. PT and APPT <2 times of normal amounts.
8. Karnofsky performance status ≥ 60.
9. The ECOG score ≤2 points.

Exclusion Criteria:

1. Pregnant (or lactating) women;
2. Uncontrolled active infection；
3. Active infection of hepatitis B virus or hepatitis C virus；
4. Human immunodeficiency virus (HIV) positive；
5. Patients with a history of myocardial infarction or severe arrhythmia within six months or those with class III or IV cardiac function according to the New York classification；
6. Any situations that the investigator believes may increase the risk of patients or interfere with the results of study.

Ages: 16 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients with hematological malignancies who were proposed for CAR-T treatment at the First Affiliated Hospital of Soochow University were enrolled in our study.
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2023-09-03 (Actual); Primary Completion 2024-09-02 (Estimated); Study Completion 2025-03-02 (Estimated)

PRIMARY OUTCOMES:
gut microbiota | From pre-lymphodepletion regimen to day 28 after CAR-T cells infusion
  diversity and composition of the gut microbiota
efficacy of CAR-T therapy | six months
  CR，PR and NR
toxicity of CAR-T therapy | six months
  Adverse events are evaluated with CTCAE V5.0

CONTACTS AND LOCATIONS:
Overall Officials: Xiaowen Tang, PhD, Study Chair — The First Affiliated Hospital of Soochow University
Locations (1):
- The First Affiliated Hospital of Soochow University, Suzhou, Jiangsu, China